CLINICAL TRIAL: NCT04277728
Title: Mismatch Between Hypoperfusion and Hypodensity on CT for the Identification of Patients With Stroke Onset Within 4.5 Hours
Brief Title: Hypoperfusion-hypodensity Mismatch for the Identification of Patients With Stroke Within 4.5 Hours
Acronym: MissPerfeCT
Status: Completed | Type: Observational
Sponsor: University Hospital Muenster (Other)
Responsible Party: Sponsor
Other Study IDs: 100001
Record Dates: First submitted 2020-02-17; First posted 2020-02-20 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: hypoperfusion-hypodensity mismatch — hypoperfusion-hypodensity mismatch on computed tomography

SUMMARY:
Intravenous thrombolysis is recommended within 4.5 hours of stroke onset. The aim of the study is to evaluate whether a hypodensity on native CT within the virtually entire area of hypoperfusion on perfusion CT, i.e. hypoperfusion-hypodensity mismatch, identifies patients within the time window of thrombolysis in a multicenter cohort. The investigators hypothesize hypoperfusion-hypodensity mismatch will identify patients ≤ 4,5 hours of symptom onset with >70% specificity and >85% positive predictive value.

ELIGIBILITY:
Inclusion Criteria:

* acute ischemic stroke
* evidence of acute intracranial vessel occlusion (any supratentorial proximal or peripheral artery of the anterior cerebral artery, middle cerebral artery or posterior cerebral artery territory) by CT hyper dense thrombus and/or CTangiography vessel occlusion and/or by ischemic perfusion deficit
* evidence for acute ischemic perfusion deficit, i.e. acute symptoms attributable to ischemic CT perfusion lesion
* complete native CT and CTperfusion performed on admission
* sufficient CT and CTperfusion quality for judgement of acute ischemic hypodensity
* known time of symptom onset.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute ischemic stroke and known time of symptom onset.
Sampling Method: Probability Sample
Enrollment: 689 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Positive predictive value of "hypoperfusion hypodensity mismatch" for the identification of patients ≤4.5 hours | on admission
Specificity of "hypoperfusion hypodensity mismatch" for the identification of patients ≤4.5 hours | on admission

CONTACTS AND LOCATIONS:
Overall Officials: Jens Minnerup, MD, Principal Investigator — University Hospital Muenster
Locations (1):
- University Hospital Münster, Münster, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sporns PB, Kemmling A, Meyer L, Krogias C, Puetz V, Thierfelder KM, Duering M, Lukas C, Kaiser D, Langner S, Brehm A, Rotkopf LT, Kunz WG, Beuker C, Heindel W, Fiehler J, Schramm P, Wiendl H, Minnerup H, Psychogios MN, Minnerup J. Computed tomography hypoperfusion-hypodensity mismatch vs. automated perfusion mismatch to identify stroke patients eligible for thrombolysis. Front Neurol. 2023 Dec 29;14:1320620. doi: 10.3389/fneur.2023.1320620. eCollection 2023. PMID 38225983
- [Derived] Sporns PB, Kemmling A, Minnerup H, Meyer L, Krogias C, Puetz V, Thierfelder K, Duering M, Kaiser D, Langner S, Massoth C, Brehm A, Rotkopf L, Kunz WG, Karch A, Fiehler J, Heindel W, Schramm P, Royl G, Wiendl H, Psychogios M, Minnerup J. CT Hypoperfusion-Hypodensity Mismatch to Identify Patients With Acute Ischemic Stroke Within 4.5 Hours of Symptom Onset. Neurology. 2021 Nov 23;97(21):e2088-e2095. doi: 10.1212/WNL.0000000000012891. Epub 2021 Oct 14. PMID 34649883